CLINICAL TRIAL: NCT00126048
Title: Randomised Controlled Trial to Evaluate the Effect of Statins on Asthma Control of Patients With Chronic Asthma
Brief Title: Trial to Evaluate the Effect of Statins on Asthma Control of Patients With Chronic Asthma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other); Asthma UK (Other); NHS Greater Clyde and Glasgow (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AR-001; Grant number:04/015; R&D:WN04RM024; Ethics committee:04/SO709/86
Record Dates: First submitted 2005-06-30; First posted 2005-08-02 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2008-09

CONDITIONS: Asthma
Keywords: Atopy; Statin; Asthma; methacholine; FEV1
MeSH Terms: conditions — Asthma | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Oral atorvastatin 40mg
  Interventions: Drug: Atorvastatin
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — 40mg tablet
  Other Names: Lipitor
  Arms: 1
Drug: Placebo — Placebo tablet
  Arms: 2

SUMMARY:
Statins are the most common type of cholesterol-lowering drugs used in clinical practice. Recent research suggests that they may also have anti-inflammatory properties, in particular by inhibition of an important inflammatory cell called a T lymphocyte. Asthma is characterised by chronic inflammation in the airways, which is thought to be regulated by the activity of T lymphocytes. The investigators have found the anti-inflammatory activity of a statin drug in an experimental model of allergic asthma and they have recently shown the beneficial effects of a statin, atorvastatin, in patients with rheumatoid arthritis. These findings demonstrate the therapeutic potential of statin-sensitive pathways in allergic airways disease. The investigators plan to perform a "proof of concept" study to determine the effectiveness of statin therapy in asthma. This randomised controlled trial will test the hypothesis that statins improve asthma control of patients with chronic asthma. The study will be a 22-week randomised controlled trial comparing the effect on asthma control of oral atorvastatin with that of a matched placebo. Each treatment will be administered for 8 weeks separated by a 6-week washout period. A total of 52 allergic asthmatic patients will be recruited to ensure that 44 patients complete the study. The investigators will examine the effect of statin therapy on lung function, symptom scores, exacerbation rates, as well as on the measurement of airway inflammation in sputum and in the blood. This study will determine the benefit of atorvastatin as an add-on therapy in asthma and establish if statins might have a role in asthma management.

DETAILED DESCRIPTION:
Study Design:

The study will be a 24-week randomised double blind crossover study comparing the effect on asthma control of oral atorvastatin therapy (40 mg daily) with that of a matched placebo. Each treatment will be administered for 8 weeks separated by a 6-week washout period and a 2-week run-in period prior to randomisation. Randomisation will be performed in sequential blocks.

Patients will be assessed on 9 visits (13 occasions, as some visits are performed over 2 days): -

Visit 1: Screening visit:

* Obtain written informed consent
* General medical history & physical examination
* Complete asthma control questionnaire
* Spirometry and reversibility testing.
* Blood sampling (35 ml) for IgE serology, lipids, liver function tests, creatinine kinase and immunological tests (including sVCAM-1, Sicam-1, Spcam, E-selectin, CRP, MCP-1, IL-6, IL-10 and TNF-alpha.).
* Eligibility check
* Issue diary card and peak flow meter
* Adjustment of asthma medication to BTS guidelines if required.

Visit 2: Baseline clinical measurements-2weeks after visit 1(or 4 weeks if any change made to baseline asthma medication [randomisation visit]):

* Complete asthma control questionnaire
* Asthma Quality of life questionnaire
* ATS score to assess severity of asthma.
* Spirometry and reversibility testing.
* Induced sputum
* Exhaled NO
* Airway responsiveness to methacholine
* Randomise patient if all criteria met.
* Issue diary card

Visits 3-9 at 2, 4, 8, 14, 16, 18 & 22 weeks after randomisation:

At each study visit the peak expiratory flow (PEF) diary will be retained and spirometry performed. Patients will record morning and evening PEF measurements and daily symptoms throughout the study. Airway responsiveness to methacholine, asthma control score, asthma quality of life questionnaire, induced sputum, exhaled NO and blood samples for immunological tests, lipids and liver functions will be performed at visits 5, 6 and 9. Pregnancy tests will be performed in all women of child-bearing age at visits 2 and 6 and subjects will be informed about adequate contraception during and for one month after the study.

If a subject is found to have elevated lipids at baseline, the study would be continued and the person referred to the appropriate specialist for further management after the study.

If a subject has an exacerbation during the wash-out phase of the study, visit 6 will be delayed until the patient has been stable for 4 weeks.

Anti-asthma drug treatment: Patients will be asked to continue on their usual anti-asthma drug therapy throughout the study.

Measurements:

Diary card recordings: asthma symptoms, PEF recordings and inhaled beta2-agonist use. PEF measurements will be undertaken by patients at home using a mini-Wright peak flow meter (Clement Clarke, Harlow, UK). The best of three measurements will be recorded twice daily (pre-treatment) in the diary. Peak flow variability will be calculated from the difference between the highest and lowest daily reading divided by the mean PEF reading multiplied by 100 (amplitude % mean). The average of 3 of the last 7 days PEF measurements before each visit will be used for analysis.

Exacerbations of asthma: Mild exacerbation defined as one of the following for 2 consecutive days: a drop in peak flow > 20% below baseline value, use of more than 3 additional puffs of reliever bronchodilator over 24 hours (excluding prophylactic puffs for exercise) as compared with baseline value or night awakening due to asthma. A severe exacerbation will be defined as any worsening of asthma control considered by the investigator or general practitioner (GP) to require a short course of oral corticosteroids/hospitalisation or decrease in morning peak flow to more than 30% below the baseline value on 2 consecutive days.

Other indices of disease severity relating to asthma: Emergency/'out of hours' visit of patients to the GP; GP visit to patient at home; GP or investigator prescribing extra treatment; Accident and emergency (A & E) department hospital attendance; hospital admission and length of stay.

Spirometry (FEV1, FVC), reversibility testing: Baseline pre-bronchodilator spirometric measurements will be recorded from the best of three attempts using a dry wedge spirometer (Vitalograph, Buckingham, UK) with measurements not varying by more than 5% or 0.2ml. Spirometric measurements will be made before and after nebulised salbutamol (2.5mg). Measurements will be performed at the same time of day (am or pm) for each patient.

Total and specific IgE: Total serum IgE and IgE to common allergens (house dust mites, grass pollen and cat dander) will be measured by enzyme immunoassay (Unicap System, Pharmacia UK Ltd, Milton Keynes, UK). Total IgE > 120 IU/L and specific IgE >0.35 IU/L are considered positive. Atopy will be defined as the presence of positive specific IgE to common allergens.

Airway responsiveness: Bronchial challenge testing with methacholine will be undertaken using Cockcroft's technique with concentrations of methacholine from 0.03 to 16 mg. A value of methacholine hyperreactivity > 16 mg/ml will be read as 16 mg/ml. Bronchial hyper-reactivity is defined as a PC20 FEV1 of < 8 mg/ml. Methacholine challenge testing will only be performed in subjects who have a baseline FEV1 of greater than 60% predicted.

Induced sputum: An ultrasonic nebuliser is filled with 3% saline and subjects inhale the nebulised solution for 7 minutes following pre-treatment with inhaled salbutamol. After this, the nebuliser is filled with 4% saline and the nebulised solution is inhaled for 7 minutes. Finally, the nebuliser is filled with 5% saline and the nebulised solution is inhaled for 7 minutes. At 5-minute intervals the inhalation is stopped to allow expectoration into a polypropylene container. The sample is kept on ice until processed for cell counts and ultra centrifugation to harvest the soluble phase of sputum. Cell counts will be performed and the supernatant stored for analysis of inflammatory mediators. The test will not be performed on subjects with an FEV1 < 1 L.

Measurement of exhaled NO: Exhaled NO will be measured on a chemiluminescence analyser (LR2149, Logan Research Ltd., Rochester, Kent). The methods used to measure exhaled NO will comply with the ATS guidelines.

Allergen-driven lymphocyte proliferative response in the blood: Peripheral blood mononuclear cells (106 cells/ml) will be cultured with autologous plasma for 3 days (mitogen or anti-CD3/28) or 7 days (recombinant Der p1 allergen) in a humidified atmosphere at 37°C/5% CO2. Proliferation will be measured by incorporation of tritiated thymidine (0.5uCi) for 16hr before harvest onto glass fibre filters and counting in a beta counter.

Other immunological tests in blood:

Luminex methodology for cytokine release & FACS technology for co-stimulator molecule expression will be employed to estimate altered cellular immune function in whole blood cultures over time.

Measurement of lipids in blood:

Cholesterol, triglycerides and HDL-cholesterol will be measured at screening and visits 5, 6 and 9.

Serum biochemistry safety checks: Blood for renal function (urea and electrolytes) and liver function tests (LFT's) will be performed before and after each treatment period and creatinine kinase will be performed at baseline.

Statistical Analysis:

Power calculations: A sample size of 44 will have 90% power to detect a difference in means of 20L/min in peak expiratory flow [PEF] (primary endpoint), assuming a standard deviation of differences of 40L/min, using a paired t-test with a 0.05 two-sided significance level. A total of 52 patients will be recruited to ensure that 44 patients complete the study.

Data processing and analysis: The primary analysis is a comparison between treatments of morning PEF. Secondary endpoints include: symptom scores, exacerbation rates, spirometry, airway responsiveness to methacholine, sputum cell counts, eNO and immunological tests in blood. The main analyses will be carried out by Normal Linear Models that include parameters for patient, period and treatment. Some variables may be unsuitable for this, in which case the within-patient treatment differences will be calculated and then analysed by either t-tests or Wilcoxon tests, as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma: This will be established symptomatically by episodic wheezing, chest tightness and/or dyspnoea and objectively confirmed by methacholine airway hyperresponsiveness or by evidence of variable airflow obstruction with an increase in FEV1 of > 12% following nebulised salbutamol (2.5mg) or diurnal peak flow variability of > 20% for 3 days in a week (with a minimum change of 60 L) during the run-in period of the study (BTS).
* Age range of 18-70 years
* Duration of asthma > 1 year and on stable medication for 4 weeks
* Receiving regular inhaled steroid treatment (≤ 1000mcg Beclomethasone equivalent daily) and no other medication for their asthma other than a short-acting bronchodilator.
* Symptomatic, defined as an asthma control questionnaire score of 1 (range 0-6) prior to randomisation or use of inhaled beta2-agonist on 5 or more days in the week before randomisation or FEV1 reversibility >12% or diurnal peak flow variability of >20% during the run-in period of the study for at least 3 days of a week.
* Stable asthma medication for at least 4 weeks prior to randomisation
* Written informed consent

Exclusion Criteria:

* Inability to demonstrate correct use of peak flow meter after instruction
* Current smokers or ex-smokers of < 1 year or ex-smokers who have smoked > 5 pack years.
* Patients with unstable asthma, defined as the presence of 1 or more of the following events in the month prior to randomisation: *emergency/'out of hours' visits of patients to the GP; *GP visit to patient at home; *A & E hospital attendance; *hospital admission.
* Patients in whom cardiovascular risk requires statin therapy
* Any known sensitivity or adverse reaction to statin, or previous evidence of myopathy or myositis plus creatinine kinase and liver function tests > x2 upper limit of normal range.
* Non-atopic asthma (specific IgE skin test negative to common allergens) [skin test wheal </= 3mm over negative control saline]
* Patients who show specific IgE sensitivity or are skin test positive to grass pollen allergen will not be recruited from mid May to the end of July (grass allergen season in the United Kingdom [UK]).
* Pregnancy/lactation. Patients who require medications known to interact with statins, such as azole antifungal agents, erythromycin, clarithromycin, cyclosporine, gemfibrozil, verapamil and amiodarone.
* Inability to fully comprehend the patient information sheet.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2005-07; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Change in PEFR | 8 weeks of treatment

SECONDARY OUTCOMES:
Change in health-related quality of life (HR-QOL) | 8 weeks
Change in asthma control score (Juniper) | 8 weeks
Change in inflammatory markers | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Neil C Thomson, FRCP, Principal Investigator — University of Glasgow
Locations (1):
- Asthma Clinical Research Centre, Level 6, Gartnavel General Hospital, Glasgow, United Kingdom

REFERENCES:
- [Background] Hothersall E, McSharry C, Thomson NC. Potential therapeutic role for statins in respiratory disease. Thorax. 2006 Aug;61(8):729-34. doi: 10.1136/thx.2005.057976. PMID 16877692
- See also: University of Glasgow Asthma Research Unit website — http://www.gla.ac.uk/departments/immunology/respiratorymedicine/
- See also: Prof Thomson's section of Glasgow Uni webpages — http://www.gla.ac.uk/stafflist?/action=person&ID=4cd4ebec8a92